CLINICAL TRIAL: NCT05762406
Title: Effect of the Use of Protective Masks on the Ability to Perform Daily Activities in Patients with Heart Failure or Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CCM1550
Record Dates: First submitted 2023-02-16; First posted 2023-03-09 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; COPD
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wearing mask (Experimental): Subjects will perform a cardiopulmonary exercise test (CPET) and a series of standardized daily activities while wearing a protective mask
  Interventions: Device: Respiratory protective mask
- Not wearing mask (No Intervention): Subjects will perform a cardiopulmonary exercise test (CPET) and a series of standardized daily activities in basal conditions

INTERVENTIONS:
Device: Respiratory protective mask — Subjects will perform a cardiopulmonary exercise test (CPET) and a series of standardized daily activities while wearing a protective mask.
  During the exercises, oxygen consumption, ventilation and other cardiorespiratory parameters will be assessed using a portable device (K5, Cosmed)
  Arms: Wearing mask

SUMMARY:
Scientific Rationale: In late 2019 and early 2020, researchers at the Wuhan Institute of Virology identified a potential new etiologic agent, called new coronavirus 2019 (nCoV-2019). Subsequently, the epidemic unleashed by this virus involved the whole world and radically changed the habits of the entire global population. Since that time, in fact, the need to contain the spread of infection through specific social distancing procedures and through the use of personal protective equipment has become compelling. The main tool was the requirement for all citizens to wear masks for airway protection. This measure has thus become in daily use for the majority of the population.

Therefore, it has become increasingly important to evaluate the impact of mask wearing on activities of daily living (ADls), both in healthy subjects, for which several evidences have already been brought, and in patients with different diseases, for which data are still insufficient to fully describe the effects.

Oxygen consumption and dyspnea during simple activities of daily living (ADLs) have already been studied in patients with heart failure (HF) and chronic obstructive pulmonary disease (COPD), and there is evidence that these subjects compared with healthy subjects perform ADLs at a higher percentage of their peak VO2 with more dyspnea. However, there are still no studies highlighting, however, the consequences of performing such activities while wearing a protective filtering facepiece particles class 2 (FFP2) mask, to date considered the most suitable to preserve the most fragile subjects from infection.

In this study, therefore, the investigators aim to asess the effects of these devices on the ability to perform ADLs by evaluating the exchanges of respiratory gases in the body during the performance of normal activities or during sleep in patients with HF or COPD compared with healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects:

* Age: 18-80 years
* Not taking cardiovascular medications
* No history of cardiovascular disease
* Normal physical examination
* Normal ECG

Inclusion criteria for subjects with HF:

* Age: 18-80 years
* New York Heart Association Class (NYHA) II to III in stable clinical condition
* Left ventricular ejection fraction (LVEF) <40%
* Ability to perform a maximal CPET

Patients with COPD:

* Age: 18-80 years
* Diagnosis of COPD stage GOLD II-III in stable clinical condition
* Absent concomitant heart disease
* Ability to perform a maximal CPET

Exclusion Criteria:

* Healthy subjects:
* Presence of concomitant diseases

Patients:

* Oxygen therapy
* Inability or contraindication to perform a maximal CPET

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of differences in VO2 expressed in mL/min/kg | 2 weeks
  Differences in oxygen consumption (VO2) in different daily activities under basal conditions and while wearing the protective mask (FFP2) in healthy subjects, heart failure patients and in COPD patients.
Evaluation of differences in ventilation expressed as L/min | 2 weeks
  Differences in ventilation (VE) in different daily activities under basal conditions and while wearing the protective mask (FFP2) in healthy subjects, heart failure patients and in COPD patients.

SECONDARY OUTCOMES:
Evaluation of differences in peripheral saturation (%) | 2 weeks
  Differences in peripheral saturation under basal conditions and while wearing the protective mask (FFP2) in healthy subjects, heart failure patients and in COPD patients..
Evaluation of differences in VE/VCO2 (slope during the exercise) | 2 weeks
  Differences in ventilation/carbon dioxide(VE/VCO2)slope under basal conditions and while wearing the protective mask (FFP2) in healthy subjects, heart failure patients and in COPD patients.
Evaluation of differences in heart rate (beats/min) | 2 weeks
  Differences in heart rate (HR) under basal conditions and while wearing the protective mask (FFP2) in healthy subjects, heart failure patients and in COPD patients.
Evaluation of differences in dyspnea (Borg scale) | 2 weeks
  Differences in dyspnea grade evaluated by Borg scale under basal conditions and while wearing the protective mask (FFP2) in healthy subjects, heart failure patients and in COPD patients.
Evaluation of differences in cardiorespiratory parameters during sleep: nocturnal apneas (number of events) | 2 weeks
  Differences in nocturnal apneas under basal conditions and while wearing the protective mask (FFP2) in healthy subjects, heart failure patients and in COPD patients..
Evaluation of differences in cardiorespiratory parameters during sleep: nocturnal hypopnea (number of events) | 2 weeks
  Differences in nocturnal hypopneas events under basal conditions and while wearing the protective mask (FFP2) in healthy subjects, heart failure patients and in COPD patients..
Evaluation of differences in nocturnal desaturation (%) | 2 weeks
  Differences in nocturnal desaturation under basal conditions and while wearing the protective mask (FFP2) in healthy subjects, heart failure patients and in COPD patients..

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cardiologico Monzino, Irccs, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No